CLINICAL TRIAL: NCT00829335
Title: Anatomical Segmental and Subsegmental Resection of the Liver for Hepatocellular Carcinoma: a New Approach by Means of Ultrasound-Guided Vessel Compression
Brief Title: Anatomical Resection of the Liver for Hepatocellular Carcinoma: a New Ultrasound Guided Approach
Status: Completed | Type: Observational
Sponsor: University of Milan (Other)
Responsible Party: GUIDO TORZILLI, University of Milan - Istituto Clinico Humanitas IRCCS
Other Study IDs: IOUS-COMP GENERAL
Record Dates: First submitted 2009-01-26; First posted 2009-01-27 (Estimated); Last update posted 2009-01-27 (Estimated); Status verified 2009-01

CONDITIONS: Hepatocellular Carcinoma
Keywords: Intraoperative ultrasound; Segmentectomy; HCC
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- HCC patients: According with the investigators previously reported selection flow-chart , patients suitable for surgical approach were those with HCC without ascites, without or with esophageal varices for which preoperative endoscopic eradication could be carried out successfully, and with serum bilirubin level lower than 1.5 mg/dl. Potential candidates to systematic segmental or subsegmental resection by IOUS-guided finger compression were considered patients with single HCC located in one or 2 adjacent segments without portal thrombosis, and anyway not demanding for its complete removal a sectional resection or wider.
  Interventions: Procedure: IOUS-GUIDED INTRAHEPATIC VESSEL COMPRESSION

INTERVENTIONS:
Procedure: IOUS-GUIDED INTRAHEPATIC VESSEL COMPRESSION — Using the IOUS, the tumor and the level targeted for compression are identified. Than, under the IOUS guidance, the surgeon compresses bilaterally the liver at the targeted position resulting in the compression of the portal pedicle feeding the tumor previously identified. This maneuver is constantly monitored in real-time just using the same microconvex probe, and it is maintained until the surface of the targeted liver area begins to discolor, at that time the first assistant marks the discolored area with the electrocautery, and the compression is released. Once the area is demarcated, liver dissection is started under intermittent Pringle's maneuver.

SUMMARY:
Anatomical resection is the gold standard approach for liver resection in patients with HCC. A new method for that by means of IOUS-guided finger compression has been devised.

DETAILED DESCRIPTION:
We herein describe a novel technique for the demarcation of the resection area by means of IOUS-guided finger compression to systematically accomplish anatomical segmental and subsegmental resections.

Using the IOUS, the tumor and the level targeted for compression are identified. Than, under the IOUS guidance, the surgeon compresses bilaterally the liver at the targeted position resulting in the compression of the portal pedicle feeding the tumor previously identified. This maneuver is constantly monitored in real-time just using the same microconvex probe, and it is maintained until the surface of the targeted liver area begins to discolor, at that time the first assistant marks the discolored area with the electrocautery, and the compression is released. Once the area is demarcated, liver dissection is started under intermittent Pringle's maneuver.

ELIGIBILITY:
Inclusion Criteria:

* Patients suitable for surgical approach carries of HCC
* Serum bilirubin level lower than 1.5 mg/dl

Exclusion Criteria:

* Presence of ascites
* Serum bilirubin level equal or higher than 1.6 mg/dl
* Conditions (size, vascular relation, or infiltration) demanding resection larger than a segmental area
* Tumor thrombus in portal or hepatic veins

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients reffered to our outpatient clinic for evaluation as carriers of HCC
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2007-01; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Technical feasibility

SECONDARY OUTCOMES:
Morbidity and mortality | 30 and 90 days

CONTACTS AND LOCATIONS:
Overall Officials: GUIDO TORZILLI, MD, PHD, Study Chair — University of Milan
Locations (1):
- Istituto Clinico Humanitas Irccs, Rozzano, MILANO, Italy

REFERENCES:
- [Background] Torzilli G, Donadon M, Marconi M, Palmisano A, Del Fabbro D, Spinelli A, Botea F, Montorsi M. Hepatectomy for stage B and stage C hepatocellular carcinoma in the Barcelona Clinic Liver Cancer classification: results of a prospective analysis. Arch Surg. 2008 Nov;143(11):1082-90. doi: 10.1001/archsurg.143.11.1082. PMID 19015467
- [Background] Torzilli G, Palmisano A, Del Fabbro D, Marconi M, Donadon M, Spinelli A, Bianchi PP, Montorsi M. Contrast-enhanced intraoperative ultrasonography during surgery for hepatocellular carcinoma in liver cirrhosis: is it useful or useless? A prospective cohort study of our experience. Ann Surg Oncol. 2007 Apr;14(4):1347-55. doi: 10.1245/s10434-006-9278-3. Epub 2007 Jan 26. PMID 17253105
- [Background] Torzilli G, Makuuchi M. Ultrasound-guided finger compression in liver subsegmentectomy for hepatocellular carcinoma. Surg Endosc. 2004 Jan;18(1):136-9. doi: 10.1007/s00464-003-9024-x. Epub 2003 Nov 21. PMID 14625736
- [Background] Torzilli G, Makuuchi M. Ultrasound-guided liver subsegmentectomy: the peculiarity of segment 4. J Am Coll Surg. 2001 Dec;193(6):706-8. doi: 10.1016/s1072-7515(01)01077-8. No abstract available. PMID 11768689
- [Background] Torzilli G, Takayama T, Hui AM, Kubota K, Harihara Y, Makuuchi M. A new technical aspect of ultrasound-guided liver surgery. Am J Surg. 1999 Oct;178(4):341-3. doi: 10.1016/s0002-9610(99)00193-2. PMID 10587196
- [Background] Torzilli G, Montorsi M, Gambetti A, Del Fabbro D, Donadon M, Bianchi P, Olivari N, Makuuchi M. Utility of the hooking technique for cases of major hepatectomy. Surg Endosc. 2005 Aug;19(8):1156-7. doi: 10.1007/s00464-004-2232-1. Epub 2005 May 26. PMID 16021373
- [Background] Torzilli G, Montorsi M, Del Fabbro D, Palmisano A, Donadon M, Makuuchi M. Ultrasonographically guided surgical approach to liver tumours involving the hepatic veins close to the caval confluence. Br J Surg. 2006 Oct;93(10):1238-46. doi: 10.1002/bjs.5321. PMID 16953487
- [Background] Torzilli G, Montorsi M, Donadon M, Palmisano A, Del Fabbro D, Gambetti A, Olivari N, Makuuchi M. "Radical but conservative" is the main goal for ultrasonography-guided liver resection: prospective validation of this approach. J Am Coll Surg. 2005 Oct;201(4):517-28. doi: 10.1016/j.jamcollsurg.2005.04.026. PMID 16183489
- [Background] Torzilli G, Donadon M, Marconi M, Botea F, Palmisano A, Del Fabbro D, Procopio F, Montorsi M. Systematic extended right posterior sectionectomy: a safe and effective alternative to right hepatectomy. Ann Surg. 2008 Apr;247(4):603-11. doi: 10.1097/SLA.0b013e31816387d7. PMID 18362622
- [Derived] Torzilli G, Procopio F, Cimino M, Del Fabbro D, Palmisano A, Donadon M, Montorsi M. Anatomical segmental and subsegmental resection of the liver for hepatocellular carcinoma: a new approach by means of ultrasound-guided vessel compression. Ann Surg. 2010 Feb;251(2):229-35. doi: 10.1097/SLA.0b013e3181b7fdcd. PMID 19838106